CLINICAL TRIAL: NCT06021613
Title: Marijuana and Acute Risk of Arrhythmia- Joint Abstinence and Exposure
Brief Title: The MARY-JANE Cannabis and Heart Rhythm Trial
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 23-39656
Record Dates: First submitted 2023-08-28; First posted 2023-09-01 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2025-06

CONDITIONS: Premature Atrial Contractions; Premature Ventricular Contractions
Keywords: Cannabis; Marijuana; Weed; Arrhythmias; Cardiac Ectopy; PACs; PVCs; Heart Rhythm
MeSH Terms: conditions — Atrial Premature Complexes; Ventricular Premature Complexes; Marijuana Abuse; Arrhythmias, Cardiac

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Case-crossover (Experimental): Participants will be randomized in two-day blocks to consume then avoid cannabis ("Start: On Cannabis") or avoid then consume cannabis ("Start: Off Cannabis"). Using an case-crossover strategy delivered by the NIH-funded, UCSF-run Eureka platform utilizing a mobile smartphone-based application, or the Mosio text messaging software for clinical research, participants will receive instructions and answer questions to help researchers and physicians understand the relationship between inhaled cannabis and heart rhythm.
  Interventions: Behavioral: Randomized instructions

INTERVENTIONS:
Behavioral: Randomized instructions — Behavioral: Start: On Cannabis- In this two-day block, participants will be instructed to consume cannabis for one day and avoid cannabis the next day. Participants will be asked to smoke or vape cannabis at least once on days they are instructed to consume cannabis.
  Behavioral: Start: Off Cannabis- In this two-day block, participants will be instructed to avoid cannabis for one day and consume cannabis the next day. Participants will be asked to smoke or vape cannabis at least once on days they are instructed to consume cannabis.

SUMMARY:
Despite recreational cannabis now being legal in 23 states, where more than 100 million Americans reside, studies on the actual health effects are limited. This study is a randomized trial, where each participant will be instructed to consume or avoid cannabis on randomly assigned days during a 14-day monitoring period. The goal of this study is to answer the question:

"Does cannabis use increase the frequency of 'early' and abnormal heart beats?"

During the 14-day period, participants will wear an external heart monitor, a glucose monitor, and a fitness tracker to track heart rhythm, glucose levels, step counts, and sleep health. Participants will use a mobile app or a text messaging service for daily instructions/reminders on cannabis use, and short surveys. The investigators ask that participants smoke or vape cannabis at least once on days they are instructed to consume cannabis. Compelling evidence of heart and other health effects would be important to the clinical care of our patients.

DETAILED DESCRIPTION:
This study is designed as a case-crossover randomized trial, where each participant will be instructed to consume or avoid inhaled cannabis on randomly assigned days during a 14-day monitoring period. Participants will be asked to smoke or vape cannabis at least once on days they are instructed to consume cannabis. Participants will also wear an external electrocardiographic (ECG) monitor, a continuous glucose monitor, and a fitness tracker for up to two weeks while utilizing a mobile application or text messaging service to receive daily instructions/reminders on cannabis use, and short surveys. The investigators will compare participant self-report of cannabis consumption, glucose monitoring, fitness levels, sleep health, and heart rhythm data in order to better understand the relationship between acute cannabis consumption and heart rhythm changes. A total of 100 participants will be enrolled at the UCSF study site.

ELIGIBILITY:
Inclusion Criteria:

1. Are age 21 or older
2. Have a smartphone
3. Are able to use the Eureka mobile application and Mosio text messaging software
4. Have inhaled cannabis in the past month and on at least four different days in the same week in the past year
5. Are willing to consume and abstain from inhaled cannabis for no more than two consecutive days as instructed over the 14-day trial period
6. Are able to participate in a location where cannabis use would not break any established laws under any jurisdiction
7. Are able to self supply cannabis throughout the study duration

Exclusion Criteria:

1. Currently pregnant or trying to get pregnant
2. Have a medical reason to avoid cannabis
3. Are unwilling to avoid all forms of cannabis consumption on days instructed to abstain from cannabis
4. Are currently taking anti-arrhythmic medications
5. Have a history of atrial fibrillation or heart failure
6. Have congenital heart disease
7. Have an implantable cardioverter-defibrillator or pacemaker
8. Have had a previous cardiac ablation procedure
9. Are currently taking insulin
10. Are unable to read or sign to provide informed consent

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-01-18 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Change in PAC and PVC frequencies | Baseline and after completion of cannabis consumption, up to 2 weeks
  Participants will be wearing a continuously recording ECG monitor for two weeks. The primary outcome will be change in premature atrial contraction (PAC) and PVC frequency due to cannabis consumption or avoidance during the monitoring period.

SECONDARY OUTCOMES:
Change in SVT episodes | Baseline and after completion of cannabis consumption, up to 2 weeks
  Participants will be wearing a continuously recording ECG monitor for two weeks. A secondary outcome will be change in supraventricular tachycardia (SVT) episodes due to cannabis consumption or avoidance during the monitoring period.
Change in VT episodes | Baseline and after completion of cannabis consumption, up to 2 weeks
  Participants will be wearing a continuously recording ECG monitor for two weeks. A secondary outcome will be change in ventricular tachycardia (VT) episodes due to cannabis consumption or avoidance during the monitoring period.
Mean daily glucose levels | 2 weeks
  Participants will be wearing a continuous glucose monitor that will record serum glucose levels. A secondary outcome will be difference in mean daily glucose levels due to cannabis consumption or avoidance during the monitoring period.
Mean step count | 2 weeks
  Participants will be wearing a fitness tracker that will record step counts. A secondary outcome will be difference in mean step counts due to cannabis consumption or avoidance during the monitoring period.
Mean sleep duration | 2 weeks
  Participants will be wearing a fitness tracker that will record sleep duration. A secondary outcome will be difference in mean sleep duration due to cannabis consumption or avoidance during the monitoring period.

CONTACTS AND LOCATIONS:
Overall Officials: Gregory M Marcus, MD, MAS, Principal Investigator — University of California, San Francisco
Locations (2):
- United States (2):
  - UCSF Medical Center at Parnassus, San Francisco, California
  - UCSF Medical Center at Mission Bay, San Francisco, California

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Colilla S, Crow A, Petkun W, Singer DE, Simon T, Liu X. Estimates of current and future incidence and prevalence of atrial fibrillation in the U.S. adult population. Am J Cardiol. 2013 Oct 15;112(8):1142-7. doi: 10.1016/j.amjcard.2013.05.063. Epub 2013 Jul 4. PMID 23831166
- [Background] Virani SS, Alonso A, Aparicio HJ, Benjamin EJ, Bittencourt MS, Callaway CW, Carson AP, Chamberlain AM, Cheng S, Delling FN, Elkind MSV, Evenson KR, Ferguson JF, Gupta DK, Khan SS, Kissela BM, Knutson KL, Lee CD, Lewis TT, Liu J, Loop MS, Lutsey PL, Ma J, Mackey J, Martin SS, Matchar DB, Mussolino ME, Navaneethan SD, Perak AM, Roth GA, Samad Z, Satou GM, Schroeder EB, Shah SH, Shay CM, Stokes A, VanWagner LB, Wang NY, Tsao CW; American Heart Association Council on Epidemiology and Prevention Statistics Committee and Stroke Statistics Subcommittee. Heart Disease and Stroke Statistics-2021 Update: A Report From the American Heart Association. Circulation. 2021 Feb 23;143(8):e254-e743. doi: 10.1161/CIR.0000000000000950. Epub 2021 Jan 27. PMID 33501848
- [Background] Dieleman JL, Cao J, Chapin A, Chen C, Li Z, Liu A, Horst C, Kaldjian A, Matyasz T, Scott KW, Bui AL, Campbell M, Duber HC, Dunn AC, Flaxman AD, Fitzmaurice C, Naghavi M, Sadat N, Shieh P, Squires E, Yeung K, Murray CJL. US Health Care Spending by Payer and Health Condition, 1996-2016. JAMA. 2020 Mar 3;323(9):863-884. doi: 10.1001/jama.2020.0734. PMID 32125402
- [Background] Marcus GM, Vittinghoff E, Whitman IR, Joyce S, Yang V, Nah G, Gerstenfeld EP, Moss JD, Lee RJ, Lee BK, Tseng ZH, Vedantham V, Olgin JE, Scheinman MM, Hsia H, Gladstone R, Fan S, Lee E, Fang C, Ogomori K, Fatch R, Hahn JA. Acute Consumption of Alcohol and Discrete Atrial Fibrillation Events. Ann Intern Med. 2021 Nov;174(11):1503-1509. doi: 10.7326/M21-0228. Epub 2021 Aug 31. PMID 34461028
- [Background] Lin AL, Nah G, Tang JJ, Vittinghoff E, Dewland TA, Marcus GM. Cannabis, cocaine, methamphetamine, and opiates increase the risk of incident atrial fibrillation. Eur Heart J. 2022 Dec 14;43(47):4933-4942. doi: 10.1093/eurheartj/ehac558. PMID 36257330
- [Background] Dewland TA, Vittinghoff E, Mandyam MC, Heckbert SR, Siscovick DS, Stein PK, Psaty BM, Sotoodehnia N, Gottdiener JS, Marcus GM. Atrial ectopy as a predictor of incident atrial fibrillation: a cohort study. Ann Intern Med. 2013 Dec 3;159(11):721-8. doi: 10.7326/0003-4819-159-11-201312030-00004. PMID 24297188
- [Background] Marcus GM, Dewland TA. Premature Atrial Contractions: A Wolf in Sheep's Clothing? J Am Coll Cardiol. 2015 Jul 21;66(3):242-244. doi: 10.1016/j.jacc.2015.04.069. No abstract available. PMID 26184617
- [Background] Dukes JW, Dewland TA, Vittinghoff E, Mandyam MC, Heckbert SR, Siscovick DS, Stein PK, Psaty BM, Sotoodehnia N, Gottdiener JS, Marcus GM. Ventricular Ectopy as a Predictor of Heart Failure and Death. J Am Coll Cardiol. 2015 Jul 14;66(2):101-9. doi: 10.1016/j.jacc.2015.04.062. PMID 26160626
- [Background] Marcus GM. Evaluation and Management of Premature Ventricular Complexes. Circulation. 2020 Apr 28;141(17):1404-1418. doi: 10.1161/CIRCULATIONAHA.119.042434. Epub 2020 Apr 27. PMID 32339046
- [Background] Marcus GM, Rosenthal DG, Nah G, Vittinghoff E, Fang C, Ogomori K, Joyce S, Yilmaz D, Yang V, Kessedjian T, Wilson E, Yang M, Chang K, Wall G, Olgin JE. Acute Effects of Coffee Consumption on Health among Ambulatory Adults. N Engl J Med. 2023 Mar 23;388(12):1092-1100. doi: 10.1056/NEJMoa2204737. PMID 36947466